CLINICAL TRIAL: NCT05844137
Title: Improving Detection and Evidence-based Care of NAFLD in Latinx and Black Patients With Type 2 Diabetes (NAFLD-DM): A Pilot Study
Brief Title: Improving Detection and Evidence-based Care of NAFLD in Latinx and Black Patients With Type 2 Diabetes
Acronym: NAFLD-DM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Duke University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Pro00113239
Record Dates: First submitted 2023-04-25; First posted 2023-05-06 (Actual); Results first posted 2024-12-27 (Actual); Last update posted 2024-12-27 (Actual); Status verified 2024-09

CONDITIONS: NAFLD; Diabetes Mellitus
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease; Diabetes Mellitus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Evidence-based care of NAFLD in T2D (Experimental): Intervention content will include: 1) NAFLD education; 2) diet/lifestyle support; 3) T2D medication management; and 4) clinically-indicated liver testing and care
  Interventions: Behavioral: NAFLD Education; Behavioral: diet/lifestyle support; Drug: T2D medication management; Diagnostic Test: clinically-indicated liver testing and care

INTERVENTIONS:
Behavioral: NAFLD Education — NAFLD Education
Behavioral: diet/lifestyle support — diet/lifestyle support
Drug: T2D medication management — T2D medication management
Diagnostic Test: clinically-indicated liver testing and care — clinically-indicated liver testing and care

SUMMARY:
The primary objective of this pilot study is to assess the feasibility and acceptability of an intervention for improved detection and evidence-based care of NAFLD in Latinx and Black patients with type 2 diabetes (T2D) in Duke University Healthcare system (DUHS). We will enroll 10-15 Latinx and 10-15 Black patients with T2D and NAFLD, based on having mildly elevated liver enzymes (ALT >/= 40 IU/mL in males, ALT >/= 31 IU/mL in females) and exclusion of other liver diseases (e.g., viral hepatitis, alcohol abuse).

Intervention content will include: 1) NAFLD education; 2)diet/lifestyle support; 3) T2D medication management; and 4) clinically-indicated liver testing and care.

Intervention feasibility will be evaluated by examining recruitment rates, retention rates, and study visit completion rates. Acceptability will be assessed by survey and through qualitative interviews. The project objectives and intervention are minimal risk. The expected risks will not exceed those of usual care.

ELIGIBILITY:
Inclusion Criteria:

* People who identify as either: Latino/Latina/Hispanic ethnicity and/or Black or African American race
* People with type 2 diabetes (T2D), as defined by ICD-10 codes E11.xx.
* Patients with elevated serum alanine aminotransferase (ALT) within Duke University Healthcare System (DUHS). Elevated ALT will be defined as having at least two ALT ≥40 IU/mL in males or ≥31 IU/mL in females in the preceding 12 months

Exclusion Criteria:

* People with hepatitis B or C infection
* People with known alcohol overuse
* People with current use of chemotherapy or other drugs known to affect liver function
* People who have not been seen by a DUHS Primary Care Physician (PCP) or Endocrinologist in the preceding year.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2023-09-18 (Actual); Primary Completion 2024-01-29 (Actual); Study Completion 2024-01-29 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Anastasia-Stefania Alexopoulos, MD, Principal Investigator — Duke University
Locations (1):
- Duke University Healthcare System, Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No
NA- IPD will not be made available to other researchers

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Evidence-based Care of NAFLD in T2D
Started | 10
Completed | 10
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: There were fewer participants than initially anticipated due to budget/resource constraints
Arm/Group | Evidence-based Care of NAFLD in T2D
Number analyzed (Participants) | 10
Age, Continuous [Mean (Standard Deviation); unit: years] | 51.1 (9.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5
  Male | 5
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 6
  Not Hispanic or Latino | 4
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 4
  White | 3
  More than one race | 0
  Unknown or Not Reported | 2
Region of Enrollment [Number; unit: participants]
  United States | 10
Non-adherence to diabetes medications [Count of Participants; unit: Participants] — Population: 9 participants were on non-insulin medications and only 1 participant was on insulin.
  Participants
    Non-insulin medications: number analyzed (Participants) | 9
    Non-insulin medications | 2
    Insulin: number analyzed (Participants) | 1
    Insulin | 1

OUTCOME MEASURES:

1. Primary Outcome: Feasibility as Measured by Recruitment Rate
Description: The Investigator will assess recruitment rates: Patients eligible and sent letter of message / Patients enrolled
Time Frame: 3 months
Population: This outcome includes all patients that were approached for recruitment either by cold call or MyChart messages.
Measure: Count of Participants; unit: Participants
Arm/Group | Evidence-based Care of NAFLD in T2D
Number analyzed (Participants) | 51
Participants
  Recruitment by Cold Call: number analyzed (Participants) | 31
  Recruitment by Cold Call | 8
  Recruitment by MyChart: number analyzed (Participants) | 20
  Recruitment by MyChart | 2

2. Primary Outcome: Feasibility as Measured by Retention Rate
Description: The team will assess retention rates: Patients enrolled / Patients completing study
Time Frame: 3months
Measure: Count of Participants; unit: Participants
Arm/Group | Evidence-based Care of NAFLD in T2D
Number analyzed (Participants) | 10
Participants | 10

3. Primary Outcome: Feasibility as Measured by Visit Completion Rate
Description: The Investigator assess visit completion rates: Total study visits completed / Total study visits scheduled
Time Frame: 3months
Population: There were 3 study visits per participant so 30 total study visits.
Measure: Number; unit: number of study visits
Units Other Than Participants: Number of Visits Scheduled
Arm/Group | Evidence-based Care of NAFLD in T2D
Number analyzed (Participants) | 10
Number analyzed (Number of Visits Scheduled) | 30
number of study visits | 30

4. Primary Outcome: Feasibility of System-level NAFLD Detection Approach
Description: Measure by the number of patients who met criteria for NAFLD after chart review / total number of potentially-eligible patients based on our EHR criteria.
Time Frame: Baseline
Population: This outcome includes potentially eligible participants identified prior to enrollment. The charts of 184 patients were reviewed and 122 patients were ultimately found to be eligible.
Measure: Number; unit: patient charts reviewed
Arm/Group | Evidence-based Care of NAFLD in T2D
Number analyzed (Participants) | 184
patient charts reviewed | 122

5. Primary Outcome: Acceptability of Intervention by Participants
Description: The Investigator will calculate the mean and standard deviation of the Treatment Acceptability and Preferences (TAP);Minimum value = 0; Maximum value = 4; Higher score is a better outcome (ie more acceptable). The Investigator define acceptable score as mean TAP ≥ 3.
Time Frame: 3months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Evidence-based Care of NAFLD in T2D
Number analyzed (Participants) | 10
score on a scale | 3.98 (0.13)

6. Secondary Outcome: Change in Self-Efficacy Measured by the Managing Chronic Diseases (SEMCD) Score
Description: The SEMCD is a 6-item scale with a total minimum value = 1; a total maximum value = 10; Higher score is a better outcome (ie greater self-efficacy). Will be measured by a change of >/=1.
Time Frame: Baseline, 3months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Evidence-based Care of NAFLD in T2D
Number analyzed (Participants) | 10
score on a scale | 0.4 (1.1)

7. Secondary Outcome: Change in Autonomy Support Measured by the Modified Health Care Climate Questionnaire (HCCQ)
Description: The HCCQ is a 5-item scale with a total minimum value = 1; a total maximum value = 5; Higher score is a better outcome (ie greater self-management)
  Will be measured by a change of >/=1 as being clinically significant.
Time Frame: Baseline, 3months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Evidence-based Care of NAFLD in T2D
Number analyzed (Participants) | 10
score on a scale | -0.1 (0.7)

8. Secondary Outcome: Change in Physical Health Quality of Living as Measured by the 12-Item Short Form Health Survey (SF-12)
Description: The SF-12 is a 5-item scale with a total minimum value = 0; a total maximum value = 100; Higher score is a better outcome (ie greater quality of life)
  Will be measured by a change of >/=10 as being clinically significant.
Time Frame: Baseline, 3months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Evidence-based Care of NAFLD in T2D
Number analyzed (Participants) | 10
score on a scale | 3.0 (3)

9. Secondary Outcome: Change in Mental Health Quality of Living as Measured by the SF-12
Description: as for outcome 8
Time Frame: Baseline, 3months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Evidence-based Care of NAFLD in T2D
Number analyzed (Participants) | 10
score on a scale | 0.5 (2.7)

10. Secondary Outcome: Change in Mean Hemoglobin A1c (HbA1c)
Description: Change of >/= 0.5% will be deemed clinically significant
Time Frame: Baseline, 3months
Population: Due to budget constraints, data were not collected.
Arm/Group | Evidence-based Care of NAFLD in T2D
Number analyzed (Participants) | 0

11. Secondary Outcome: Change in Mean Alanine Aminotransferase (ALT) Level
Description: Change of >/= 5 IU/mL will be deemed clinically significant.
Time Frame: Baseline, 3months
Population: Due to budget constraints, data were not collected.
Arm/Group | Evidence-based Care of NAFLD in T2D
Number analyzed (Participants) | 0

12. Secondary Outcome: Number of Participants With Changes to Medications During the Study Period Measured by Chart Review
Time Frame: baseline, 3 months
Measure: Count of Participants; unit: Participants
Arm/Group | Evidence-based Care of NAFLD in T2D
Number analyzed (Participants) | 10
Participants | 5

13. Secondary Outcome: Number of Participants in Whom Clinically-indicated Tests Were Ordered (e.g. Labs, Referral, Imaging).
Time Frame: baseline, 3 months
Measure: Count of Participants; unit: Participants
Arm/Group | Evidence-based Care of NAFLD in T2D
Number analyzed (Participants) | 10
Participants
  Labs Ordered | 7
  Imaging Ordered | 2
  Hepatology referral placed | 1

ADVERSE EVENTS:
Time Frame: 3 months
Arm/Group | Evidence-based Care of NAFLD in T2D
All-Cause Mortality (participants affected / at risk) | 0/10
Serious Adverse Events (participants affected / at risk) | 0/10
Other Adverse Events (participants affected / at risk) | 0/10

LIMITATIONS AND CAVEATS:
Due to resources constraints, we did not achieve our target number of participants. We did not conduct effect size calculations or inferential statistics due to the small sample size and pilot nature of this study. Further, larger studies will be necessary to examine the effectiveness of this approach - across broader racial and ethnic identities - and to determine the effectiveness of this intervention (versus usual care) on clinically-relevant outcomes.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (3):
  • Study Protocol (2024-05-31): https://cdn.clinicaltrials.gov/large-docs/37/NCT05844137/Prot_001.pdf
  • Statistical Analysis Plan (2024-05-31): https://cdn.clinicaltrials.gov/large-docs/37/NCT05844137/SAP_002.pdf
  • Informed Consent Form (2023-05-18): https://cdn.clinicaltrials.gov/large-docs/37/NCT05844137/ICF_000.pdf